CLINICAL TRIAL: NCT06132880
Title: Effects of Human Urinary Kallidinogenase on Early Improvement and Functional Outcomes in Acute Ischemic Stroke: a Multicenter, Randomized, Open Label, Blinded-endpoint, Controlled Study (TK-SPEED)
Brief Title: Effects of Human Urinary Kallidinogenase on Early Improvement and Functional Outcomes in Acute Ischemic Stroke (TK-SPEED)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Collaborators: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KLK-S024
Record Dates: First submitted 2023-11-08; First posted 2023-11-15 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Acute Ischemic Stroke; Functional Outcomes
Keywords: Acute Ischemic Stroke; Functional Outcomes; Early cerebral perfusion; Human Urinary Kallidinogenase
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intravenous injections of urinary kallidinogenase (0.15 peptide nucleic acids (PNA) in 0.9% NaCl) intravenous drip quaquedie (QD) for 10 days.
  Interventions: Drug: Human Urinary Kallidinogenase; Other: Clinical Routine Treatment
- Control group (Other): Conventional therapy of acute ischemic stroke after based on Chinese guidelines.
  Interventions: Other: Clinical Routine Treatment

INTERVENTIONS:
Drug: Human Urinary Kallidinogenase — Intravenous injections of urinary kallidinogenase (0.15 peptide nucleic acids (PNA) in 0.9% NaCl) intravenous drip QD for 10 days.
  Arms: Intervention group
Other: Clinical Routine Treatment — Conventional therapy of acute ischemic stroke after based on Chinese guidelines

SUMMARY:
The primary purpose of this trial is to evaluate the effects of Human Urinary Kallidinogenase on improvement of neurological outcome, and early cerebral perfusion in acute ischemic stroke.

DETAILED DESCRIPTION:
This is a multicentre, randomized, open label, blinded-endpoint trial that aims to investigate the effects of Human Urinary Kallidinogenase treatment on neurological outcomes, early cerebral perfusion in patients with acute anterior circulation ischemic stroke. Patients in intervention group will be given 0.15 peptide nucleic acids (PNA) Human Urinary Kallidinogenase concentrated solution for intravenous injection once a day for 10 days continuously, and those in the control group will be given conventional therapy. Both groups of patients will be on standard stroke care. In this study, patients who were eligible to the inclusion criteria and ineligible to the exclusion criteria will be randomly assigned into two groups by a 1:1 ratio after the informed consent form (ICF) was received. The total sample size will be 540. All patients will be followed up for 90 days. The primary outcome is the proportion of modified Rankin Scale 0-2. Besides, the investigators aimed to use computed tomography perfusion (CTP) evaluate the differences of ischemic penumbra volume and regional cerebral blood flow (rCBF) before and after treatment between intervention group and control group.

Furthermore, this study adopts adaptive design, prospectively stating interim analyses with specified stopping rules, which allow for the possibility of the study to terminate early based on either determination of study success or of the futility to continue further enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 80 years of age;
2. Diagnosis of anterior circulation acute ischemic stroke;
3. Within 48 hours of symptoms onset;
4. modified Rankin Scale (mRS) score≤1 before this event;
5. 5≤NIHSS≤20 at screening;
6. The availability of informed consent.

Exclusion Criteria:

1. Patients who have already or are going to receive intravenous thrombolytic/mechanical thrombectomy therapy after onset;
2. Patients with severe consciousness disorder, NIHSS 1a consciousness level score≥2;
3. Patients with limited limb mobility such as fractures and claudication upon admission;
4. Patients who have already or are going to receive Edaravone injection, Edaravone and DeKanol concentrated solution for injection, Butylphthalide and sodium chloride injection or Butylphthalide soft capsules after onset;
5. Hypotensive (systolic blood pressure <90 mmHg or diastolic blood pressure<60 mmHg) on admission;
6. History of severe drug or food allergy, allergy or intolerance to Human Urinary Kallidinogenase;
7. Patients who have been on angiotensin-converting enzyme inhibitor (ACEI) drugs and within 5 half-lives (according to the specific drug instructions) before initiate Human Urinary Kallidinogenase treatment;
8. Pregnancy, lactation, or planned pregnancy within 90 days;
9. Patients with severe renal failure or impairment (eGFR<30ml/min/1.73m2) at screening;
10. Severe hepatic dysfunction, elevation of alanine aminotransferase (ALT) or aspartate aminotransferase (AST) (more than 2.5 times of upper limit of normal value), other liver diseases such as acute and chronic hepatitis, cirrhosis, etc;
11. Patients with heart failure (NYHA class III or IV), unstable angina pectoris, acute myocardial infarction, severe arrhythmia, and degree II and III cardiac conduction obstruction within 6 months prior to randomization;
12. Heavy drinking in the three months before screening, drinking≥5 standard drinks per day (1 standard drink is equivalent to120ml wine, 360ml beer or 45ml liquor);
13. Drug Abuse or addiction in the past year;
14. Patients with a malignant tumor, severe systemic diseases, or estimated survival time <90 days;
15. Patients with severe mental disorders or dementia unable to complete the informed consent and follow-up;
16. Have participated in another interventional clinical study within 30 days before randomization or are participating in another interventional clinical study;
17. Other cases unsuitable for this clinical study assessed by researcher.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2023-12-14 (Estimated); Primary Completion 2026-08-28 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with modified Rankin Scale (mRS) 0-2 at day 90 | 90 days
  The proportion of patients with modified Rankin Scale (mRS) 0-2 at day 90. mRS scores range from 0 to 6. 0=no symptoms,1 = symptoms without clinically significant disability,2 = slight disability,3 = moderate disability,4 = moderately severe disability,5 = severe disability; and 6 = death.

SECONDARY OUTCOMES:
Change of Tmax>6s volume | 5 days
  Change of Tmax>6s volume on CTP from baseline to 5 days after treatment
Change of rCBF in Tmax>6s area | 5 days
  Change of rCBF in Tmax>6s area on CTP from baseline to 5 days after treatment
Ordinal distribution of modified Rankin Scale (mRS) at day 90 | 90 days
  Ordinal distribution of modified Rankin Scale (mRS) at day 90. mRS scores range from 0 to 6. 0=no symptoms,1 = symptoms without clinically significant disability,2 = slight disability,3 = moderate disability,4 = moderately severe disability,5 = severe disability; and 6 = death.
The proportion of patients with modified Rankin Scale (mRS) 0-1 at day 90 | 90 days
  The proportion of patients with modified Rankin Scale (mRS) 0-1 at day 90. mRS scores range from 0 to 6. 0=no symptoms,1 = symptoms without clinically significant disability,2 = slight disability,3 = moderate disability,4 = moderately severe disability,5 = severe disability; and 6 = death.
Change of National Institute of Health stroke Scale (NIHSS) score at day 5 after treatment. | 5 days
  Change of National Institute of Health stroke Scale (NIHSS) score from baseline to 5 days after treatment. NIHSS ranges from 0 to 42, a low value represents a better outcome.
Change of National Institute of Health stroke scale (NIHSS) score at day 10 after treatment. | 10 days
  Change of National Institute of Health stroke scale (NIHSS) score from baseline to 10 days after treatment. NIHSS ranges from 0 to 42, a low value represents a better outcome.

OTHER OUTCOMES:
Change of regional cerebral blood volume (rCBV) in Tmax>6s area | 5 days
  Change of regional cerebral blood volume (rCBV) in Tmax>6s area on CTP from baseline to 5 days after treatment
Change of mean transit time (MTT) in Tmax>6s area | 5 days
  Change of mean transit time (MTT) in Tmax>6s area on CTP from baseline to 5 days after treatment
Change of Tmax>4s volume | 5 days
  Change of Tmax>4s volume on CTP from baseline to 5 days after treatment
Change of Tmax>8s volume | 5 days
  Change of Tmax>8s volume on CTP from baseline to 5 days after treatment
Change of Tmax>10s volume | 5 days
  Change of Tmax>10s volume on CTP from baseline to 5 days after treatment
Change of National Institute of Health stroke scale (NIHSS) score at day 3 after treatment. | 3 days
  Change of National Institute of Health stroke scale (NIHSS) score from baseline to 3 days after treatment. NIHSS ranges from 0 to 42, a low value represents a better outcome.
Stroke recurrence rate | 90 days
  Stroke recurrence rate within 90 days
Infarct core volume | 5 days
  Infarct core volume at 5 days after treatment on diffusion weighted imaging (DWI)
Mini-Mental State Examination (MMSE) at day 90. | 90 days
  Mini-mental State Examination（MMSE）at day 90. The MMSE uses a 0-30 score scale which effected by age and education experience. Cognitive impairment is diagnosed when MMSE ≤17 for illiteracy，MMSE ≤20 for those who take less than 6-years primary education，MMSE ≤24 for those have at least a middle school education.
Montreal Cognitive Assessment (MoCA) at day 90. | 90 days
  Montreal Cognitive Assessment (MoCA) at day 90. The MoCA uses a 0-30 score scale and defines impairment as follows: score of 18-25=mild,10-17=moderate and <10 =severe.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Wu, Study Chair — Beijing Tsinghua Changgeng Hospital; Zunjing Liu, Study Chair — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: No